CLINICAL TRIAL: NCT01353976
Title: A Multi-Center, Randomized, Double-Blind, Vehicle Controlled, Parallel Group Comparison Study of the Safety and Efficacy of Econazole Nitrate Foam 1% and Foam Vehicle in Subjects With Interdigital Tinea Pedis
Brief Title: Safety and Efficacy of Econazole Nitrate Foam 1% in Subjects With Tinea Pedis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AmDerma (Industry)
Collaborators: AmDerma Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 079-2951-302
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2012-12

CONDITIONS: Tinea Pedis; Athlete's Foot
Keywords: Econazole Nitrate; Foam; Quinnova; Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Econazole Nitrate Foam 1% (Experimental): Study medication
  Interventions: Drug: Econazole Nitrate Foam 1%
- Vehicle Foam (Placebo Comparator): Placebo medication
  Interventions: Other: Vehicle Foam

INTERVENTIONS:
Drug: Econazole Nitrate Foam 1% — Econazole Nitrate Foam 1% applied once a day for 4 weeks
  Arms: Econazole Nitrate Foam 1%
Other: Vehicle Foam — Vehicle foam applied once a day for 4 weeks
  Arms: Vehicle Foam

SUMMARY:
This is a study of the safety and efficacy of topical Econazole Nitrate Foam 1% and the foam vehicle in subjects with interdigital tinea pedis (athlete's foot between the toes). This is a 6 week study which has a 4 week treatment period and a 2 week follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 12 years of age and of either sex.
* Have a clinical diagnosis of interdigital tinea pedis involving at least2 web spaces in total which extends no more than approximately 1 inch proximal to the web spaces or metatarsophalangeal joints with at least i) moderate scaling and ii) mild erythema defined as a Grade 2 and Grade 1, respectively on the Grading of Signs and Symptoms at baseline.
* Be willing and able to give informed consent/assent or have their parent/guardian do so, if applicable.
* Be willing and able to use the assigned study medication as directed and to commit to all follow-up visits for the duration of the study.
* Have microscopic evidence (positive KOH) of the presence of fungi. Evaluable subjects must have a positive KOH and a fungal culture positive for a dermatophyte in the skin scrapings taken at the Baseline Visit. Subjects with a positive KOH may be entered into the study pending the results of the fungal culture.
* Be in good health and free of any disease or physical condition which might, in the Investigator's opinion, expose the subject to an unacceptable risk by study participation.
* Females must be non-pregnant (confirmed by a negative urine pregnancy test at baseline), non-lactating and not intending to become pregnant during the course of the study.

Exclusion Criteria:

* Is pregnant, nursing or planning a pregnancy during the study.
* Has used topical antifungals or topical corticosteroids on the feet within 30 days prior to the start of the study.
* Has received systemic antifungal therapy within 12 weeks prior to the start of the study medication.
* Has used systemic antibacterials or systemic corticosteroids within 30 days prior to the start of the study. Systemic corticosteroids do not include intranasal, inhaled, and ophthalmic corticosteroids used for the management of allergies, pulmonary disorders or other conditions.
* Has a history of uncontrolled diabetes mellitus or is immunocompromised (due to disease, e.g., HIV, or medications).
* Has concurrent tinea infection e.g. tinea versicolor, tinea cruris, moccasin-type tinea pedis, etc. (in the opinion of the Investigator).
* Onychomycosis, involving ≥ 20% of the area of either great toenail or involvement of more than five toenails in total.
* Has any other skin disease which might interfere with the evaluation of tinea pedis.
* Is currently enrolled in an investigational drug or device study.
* Has received an investigational drug or treatment with an investigational device within 30 days prior to entering this study.
* Is unreliable, including subjects with a history of drug or alcohol abuse.
* Has known hypersensitivity to any of the components of the study medications.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Piacquadio, MD, Study Director — Therapeutics, Inc.
Locations (7):
- United States (7):
  - Francisco Flores, MD, Miramar, Florida
  - Daniel M. Stewart, DO, Clinton Township, Michigan
  - Cyaandi Dove, DPM, Las Vegas, Nevada
  - Robert S. Haber, MD, South Euclid, Ohio
  - Cynthia Strout, MD, Mt. Pleasant, South Carolina
  - Michael H. Gold, MD, Nashville, Tennessee
  - Jeffrey Adelglass, MD, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Econazole Nitrate Foam 1% | Vehicle Foam
Started | 130 | 134
Completed | 82 | 83
Not Completed | 48 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Econazole Nitrate Foam 1% | Vehicle Foam | Total
Number analyzed (Participants) | 130 | 134 | 264
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 121 | 125 | 246
  >=65 years | 5 | 6 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 41.7 (12.48) | 42.5 (12.85) | 42.1 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 56 | 101
  Male | 85 | 78 | 163
Region of Enrollment [Number; unit: participants]
  United States | 91 | 92 | 183
  Dominican Republic | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Complete Cure
Description: Complete Cure is defined as a negative KOH and negative fungal culture and no evidence of clinical disease as indicated by scores of 0 (none) for each sign and symptom at Day 43.
Time Frame: Day 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Econazole Nitrate Foam 1% | Vehicle Foam
Number analyzed (Participants) | 82 | 83
Participants
  No | 63 | 81
  Yes | 19 | 2

2. Secondary Outcome: Effective Treatment
Description: Effective Treatment defined as negative KOH, negative fungal culture, no or mild (a score of 0 or 1) erythema and/or scaling with all other signs or symptoms being absent (score = 0) at Day 43.
Time Frame: Day 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Econazole Nitrate Foam 1% | Vehicle Foam
Number analyzed (Participants) | 82 | 83
Participants
  No | 42 | 74
  Yes | 40 | 9

3. Secondary Outcome: Mycological Cure
Description: Mycological Cure defined as negative KOH and negative culture at Day 43.
Time Frame: Day 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Econazole Nitrate Foam 1% | Vehicle Foam
Number analyzed (Participants) | 82 | 83
Participants
  No | 26 | 70
  Yes | 56 | 13

ADVERSE EVENTS:
Arm/Group | Econazole Nitrate Foam 1% | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 0/130 | 1/134
Other Adverse Events (participants affected / at risk) | 17/130 | 16/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Econazole Nitrate Foam 1% (N=130) | Vehicle Foam (N=134)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Econazole Nitrate Foam 1% (N=130) | Vehicle Foam (N=134)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application Site Dermatitis (General disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Sinusitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 6 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No